CLINICAL TRIAL: NCT05977426
Title: The Effects of Reiki on Menopausal Symptoms and Depression Levels in the Postmenopausal Period: A Randomized Clinical Trial
Brief Title: The Effects of Reiki on Menopausal Symptoms and Depression Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra SABANCI BARANSEL, Assit. Prof, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/4577
Record Dates: First submitted 2023-07-25; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Therapeutic Touch; Menopausal Symptoms
Keywords: Reiki; menopause; menopausal symptoms; depression
MeSH Terms: conditions — Depression | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial
Who Masked: Participant
Masking Description: This study was designed as a randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): A sociodemographic questionnaire including questions about age, last menstrual period, education level and income level, Menopause Rating Scale (MRS), Beck Depression Inventory (BDI) were utilized for the collection of research data. And a question investigating the level of being affected by menopause complaints. The question investigating the level of being affected by menopause is: "At which level do menopause complaints affect you?". Women answered this question on a scale of 0 (very little/very slightly) to 10 (extreme/very much). Data were collected from women who applied to the FHC for general healthcare services after receiving service. Women in the experimental group received Reiki once a week for four weeks. No initiative was applied to the pregnant women in the control group. Each session lasted 30-40 minutes. Four weeks after the data collection tools used in the research were filled in as a pre-test, post-test data were obtained with the same measurement tools.
  Interventions: Other: Reiki
- Routine checks (No Intervention): The researchers applied no initiative to the control group, and the women in the control group solely had the routine checks. The women in the control group filled out all pretest forms(A sociodemographic questionnaire including questions about age, last menstrual period, education level and income level, Menopause Rating Scale (MRS), Beck Depression Inventory (BDI)). The post-test forms (MRS, BDI) were re-administered 4 weeks later to women who did not receive any intervention.

INTERVENTIONS:
Other: Reiki — In the study, women received four Reiki sessions once a week for four weeks from the researchers with Usuı Shiki Ryoho Reiki 1
  Arms: Reiki

SUMMARY:
Objective: This study was conducted to determine the effects of Reiki applied to women in the postmenopausal period on menopausal symptoms and depression levels.

Methodology:This randomized controlled study was conducted with postmenopausal women registered in a family health center in eastern Türkiye. The sample of the study consisted of 82 women, 41 in the Reiki group and 41 in the control group. While four sessions of Reiki were applied to the women in the Reiki group, once a week for 4 weeks, no intervention was applied to the control group. Menopause Rating Scale (MRS) and Beck Depression Inventory (BDI) were used to collect data.

DETAILED DESCRIPTION:
Design This study was designed as a randomized controlled trial in which participants were randomly assigned to Reiki or control groups.

Location and time The study was conducted with postmenopausal women registered at a Family Health Center (FHC) located in the center of a province in eastern Türkiye between May 2023 and July 2023. The center is a primary healthcare institution that provides general healthcare services and reproductive healthcare services (such as family planning, education, and counseling). There is no application specific to the menopausal period in the center. This center was randomly selected considering its socioeconomic level, proximity to the city center, and the number of women registered in the center. The center serves approximately 15.000 individuals, of which approximately 5100 are women. In addition, there was a quiet and calm hall in the center where Reiki could be practiced.

Population and sample of the study The population of the study consisted of postmenopausal women registered to the determined FHC. Women who applied to the FHC for any reason, agreed to participate voluntarily, and met the inclusion criteria were included in the study. The criteria for inclusion in the study were as follows: Those who were between the ages of 45-55, did not have hearing problems, did not have any psychiatric diseases, were in a natural menopause period, and did not take hormone replacement therapy.

A web-based software was used to determine the sample size. Priori-power analysis was performed to estimate the appropriate sample size. In the literature, the mean score of menopausal symptoms, which is the primary result of the study, was found to be 16.6 (standard deviation 8.9). The sample size was calculated as 41 for each group (41 Reiki group, 41 control group), assuming a 5% error level, bidirectional significance level, 95% confidence interval, 80% representation of the population, and assuming to create a decrease in the post-intervention menopausal symptoms mean score by 5 points.

To reach the sample size, 140 women were evaluated in terms of eligibility criteria. 47 women who did not meet the inclusion criteria and 19 women who refused to participate in the study were excluded from the study. 7 out of 50 women included in the Reiki group were excluded from the study because they did not continue the sessions after the second Reiki session. Seven of the 53 women included in the control group were excluded from the study because they did not want to continue the study. The research was completed with a total of 82 women, 41 of them in the Reiki group and 41 of them in the control group.

Randomization The allocation of women to the Reiki and control groups in the study was done by simple randomization. For randomization, using the random number generation method available on the random.org site, numbers in which the numbers 1 and 2 are randomly sorted were created in the system. Women who accepted to participate in the study and met the inclusion criteria were randomly assigned to number 1 or 2 according to the order of arrival at the FHC. Which number would be the Reiki or control group was determined by drawing lots before starting the study. Number 1 formed the Reiki group, number 2 formed the control group. The same method was continued until the women in the Reiki and control groups reached the sample size.

Data collection tools In the study, data were collected with a sociodemographic questionnaire including questions about age, last menstrual period, education level and income level, Menopause Rating Scale (MRS), Beck Depression Inventory (BDI), and a question investigating the level of being affected by menopause complaints. The question investigating the level of being affected by menopause is: "At which level do menopause complaints affect you?". Women answered this question on a scale of 0 (very little/very slightly) to 10 (extreme/very much).

The Menopause Rating Scale (MRS) was developed to assess the severity of menopausal symptoms. The Turkish validity and reliability of the scale was performed in 2005. The scale consists of 11 items and 3 subscales. These 3 subscales are called somato-vegetative complaints (such as night sweating and hot flush), psychological complaints (such as anxiety and depression), and urogenital complaints (such as urethral syndrome and vaginal dryness). The scale is in the form of a 5-point Likert type and each item is graded between zero (no complaints) and four (severe symptoms) points. The total score that can be obtained from the scale varies between 0-44 points. An increase in the total score obtained from the scale indicates that the menopausal complaints experienced are intensified. The Cronbach's alpha reliability coefficient of the scale was calculated as 0.84.

Beck Depression Inventory (BDI) is used to have information about depressive symptoms and attitudes by evaluating the findings of emotional, cognitive, and motivational symptoms that can be seen in depression. The Turkish validity and reliability study of the inventory was carried out. Depressive symptoms and attitudes were collected under 21 headings (moodiness, pessimism, sense of failure, joylessness, sense of guilt, sense of punishment, self-blame, suicidal ideation, desire to cry, level of irritability, social loneliness, indecision, change in body image, inability to work, sleep disorder, fatigue, loss of appetite, weight loss, somatic complaints, and loss of libido). Each item is scored between 0 (not at all) and 3 (severe) according to the severity of the displayed behavior. The lowest score that can be obtained from the inventory is 0, and the highest score is 63. A high total score indicates a high level of depression severity. The Cronbach's alpha reliability coefficient of the scale was determined as 0.80.

Data collection In the study, data were collected from women who applied to the FHC for general healthcare services after receiving service. After being informed about the research by the researcher ESB, data collection tools were applied to the volunteer women in a hall in the FHC by face-to-face interview method. Four weeks after the data collection tools used in the research were filled in as a pre-test, post-test data were obtained with the same measurement tools.

Intervention The Reiki intervention was administered free of charge by the ESB from researchers holding a Usui Shiki Ryoho Reiki 1 (Degree 1) in the study. The researcher received training and certification in Reiki techniques before starting the study. After completing the training program, the researcher applied Reiki to the Reiki group once a week for 4 weeks. The sessions were held individually in a hall in the ASM, taking into account the times available to the women in the sample. Each session lasted 30-40 minutes. The Reiki application in the study was based on the First Degree Reiki (Reiki I) protocol. In Reiki I, the "aura attunement" between the practitioner and the person provides healing by touching or holding the hands a few cm above the body. The following sequence is generally applied in the Reiki protocol. 1. Before starting Reiki, the jewelry on the practitioner and the participant is removed. 2. The person sits or lies down in a comfortable position. The arms and legs remain open so that they do not touch each other. 3. Keeping the practitioner's fingers in a comfortable position, energy is sent to each chakra or area on the body for 3-5 minutes. 6. Hands are washed. In addition to the general protocol of reiki, the practitioner preferred a quiet room and dimmed the light of the room to prevent distraction and practiced in a dim environment. No intervention was applied to the control group by the researcher. Women in the control group received the service they needed from ASM.

ELIGIBILITY:
Inclusion Criteria:

* who were between the ages of 45-55,
* did not have hearing problems,
* did not have any psychiatric diseases,
* were in a natural menopause period,
* did not take hormone replacement therapy.

Exclusion Criteria:

* having a diagnosis of any psychiatric illness

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women between the ages of 45-55 years
Enrollment: 82 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-23 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | Change from menopause symptoms levels at 4 weeks
  The Menopause Rating Scale (MRS) assess the severity of menopausal symptoms. The scale consists of 11 items and 3 subscales. These 3 subscales are called somato-vegetative complaints (such as night sweating and hot flush), psychological complaints (such as anxiety and depression), and urogenital complaints (such as urethral syndrome and vaginal dryness). The scale is in the form of a 5-point Likert type and each item is graded between zero (no complaints) and four (severe symptoms) points. The total score that can be obtained from the scale varies between 0-44 points. An increase in the total score obtained from the scale indicates that the menopausal complaints experienced are intensified.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Change from depression levels at 4 weeks
  Beck Depression Inventory (BDI) is used to have information about depressive symptoms and attitudes by evaluating the findings of emotional, cognitive, and motivational symptoms that can be seen in depression. Depressive symptoms and attitudes were collected under 21 headings (moodiness, pessimism, sense of failure, joylessness, sense of guilt, sense of punishment, self-blame, suicidal ideation, desire to cry, level of irritability, social loneliness, indecision, change in body image, inability to work, sleep disorder, fatigue, loss of appetite, weight loss, somatic complaints, and loss of libido). Each item is scored between 0 (not at all) and 3 (severe) according to the severity of the displayed behavior. The lowest score that can be obtained from the inventory is 0, and the highest score is 63. A high total score indicates a high level of depression severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Sabanci Baransel, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No